CLINICAL TRIAL: NCT04201574
Title: A Phase 1/2a, Randomized, Double-Masked, Vehicle-Controlled Study Evaluating the Safety and Exploratory Activity of Two Concentrations of ALY688 Ophthalmic Solution in Subjects With Dry Eye Disease
Brief Title: Phase 1/2a Safety and Efficacy of ALY688 Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allysta Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALY688-201
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle Ophthalmic Solution
  Interventions: Drug: Vehicle
- ALY688 0.1% (Experimental): ALY688 0.1% Ophthalmic Solution
  Interventions: Drug: ALY688 0.1%
- ALY688 0.4% (Experimental): ALY688 0.4%Ophthalmic Solution
  Interventions: Drug: ALY688 0.4%

INTERVENTIONS:
Drug: ALY688 0.1% — ALY688 0.1% Ophthalmic Solution
  Other Names: ALY688 Ophthalmic
  Arms: ALY688 0.1%
Drug: ALY688 0.4% — ALY688 0.4% Ophthalmic Solution
  Other Names: ALY688 Ophthalmic
  Arms: ALY688 0.4%
Drug: Vehicle — Vehicle Ophthalmic Solution
  Other Names: placebo
  Arms: Vehicle

SUMMARY:
Clinical Trial Evaluating the Safety and Tolerability of ALY688 in Subjects with Dry Eye Disease

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked Phase 1/2a trial designed to evaluate the safety and tolerability of ALY688 Ophthalmic Solution in subjects with moderate to mildly severe dry eye for 8 weeks with 6 scheduled clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Dry eye disease for > 3 months meeting specific sign and symptom criteria
* Best correct visual acuity of +0.6 logMAR or better
* Willing to sign informed consent and attend study visits
* Willing to comply with contraception requirements

Exclusion Criteria:

* Unable to meet specific sign and symptom criteria
* Signs of ophthalmic allergic, inflammatory or infectious conditions
* Use of contact lenses
* Anatomic abnormalities preventing accurate study assessments
* Use of medications that influence eye dryness
* Recent ophthalmic surgery
* Unwilling to suspend current treatments for dry eye disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, MD, Study Director — Allysta Pharmaceutical
Locations (1):
- Allysta Pharmaceuticals, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 investigational sites in the United States
Groups:
- Vehicle Ophthalmic Solution: Vehicle Ophthalmic Solution (control arm)
- ALY688 Ophthalmic Solution 0.1%: ALY688 Ophthalmic Solution Concentration 1
- ALY688 Ophthalmic Solution 0.4%: ALY688 Ophthalmic Solution Concentration 2
Period: Overall Study
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Started | 46 | 46 | 46
Completed | 46 | 46 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: mITT Population
Groups:
- Vehicle Ophthalmic Solution: Vehicle Ophthalmic Solution (control)
- Total: Total of all reporting groups
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4% | Total
Number analyzed (Participants) | 46 | 46 | 46 | 138
Age, Continuous [Median (Full Range); unit: years] | 62.0 [23 to 86] | 63.0 [40 to 84] | 64.5 [40 to 83] | 63.0 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 36 | 102
  Male | 14 | 12 | 10 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 11 | 11 | 34
  White | 31 | 34 | 33 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 46 | 46 | 138
Eye Dryness Score [Mean (Standard Deviation); unit: units on a scale] — Eye Dryness Score using a 0- to 100-unit visual analog scale, with 0 being better and 100 being worse
  units on a scale | 66.39 (14.353) | 67.28 (12.715) | 64.48 (11.407) | 66.05 (12.841)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Subjects reporting any treatment-emergent adverse events
Time Frame: 8 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
Participants | 13 | 15 | 10

2. Primary Outcome: Eye Dryness Score (7-Day Average)
Description: Mean change from baseline in eye dryness score (7-day average) using a 0- to 100-unit visual analog scale, with 0 being better and 100 being worse
Time Frame: 8 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | ALY688 0.1% | ALY688 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale | -6.48 (2.62) | -5.66 (2.62) | -11.14 (2.64)

3. Primary Outcome: Corneal Fluorescein Staining
Description: Mean change from baseline in zonal corneal fluorescein staining score in study eye using a 0- to 4-unit clinical grading scale, with 0 being better and 4 being worse
Time Frame: 8 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale
  Zone 1 | -0.33 (0.10) | -0.37 (0.10) | -0.51 (0.10)
  Zone 2 | -0.31 (0.08) | -0.21 (0.08) | -0.36 (0.08)
  Zone 3 | -0.44 (0.09) | -0.45 (0.09) | -0.51 (0.09)
  Zone 4 | -0.40 (0.12) | -0.43 (0.11) | -0.67 (0.12)
  Zone 5 | -0.54 (0.13) | -0.42 (0.13) | -0.81 (0.13)

4. Secondary Outcome: Ocular Discomfort Score by Visual Analog Scale
Description: Mean change from baseline in ocular discomfort score of 7-day average using a 0- to 100-unit visual analog scale, with 0 being better and 100 being worse
Time Frame: 8 weeks
Population: Modified Intent-to-Treat (mITT) Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale | -8.19 (16.314) | -4.47 (17.310) | -8.62 (23.926)

5. Secondary Outcome: Symptom Assessment in Dry Eye (SAnDE) Score Assessment
Description: Mean change from baseline in Symptom Assessment in Dry Eye global symptom score on a 0- to 100-unit visual analog scale, with 0 being better and 100 being worse. Global symptom score is calculated as the square root of the frequency score time the severity score per visit
Time Frame: 8 weeks
Population: mITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale | -13.76 (19.247) | -6.76 (16.840) | -15.48 (25.219)

6. Secondary Outcome: Conjunctival Lissamine Green Staining
Description: Mean change from baseline in zonal conjunctival lissamine green staining in study eye using a 0- to 4-unit clinical grading scale, with 0 being better and 4 being worse
Time Frame: 8 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale
  Zone 1 | 0.12 (0.10) | -0.13 (0.10) | -0.18 (0.10)
  Zone 2 | -0.04 (0.11) | -0.25 (0.11) | -0.31 (0.11)
  Zone 3 | 0.02 (0.12) | -0.15 (0.11) | -0.26 (0.12)
  Zone 4 | -0.22 (0.11) | -0.37 (0.11) | -0.22 (0.11)
  Zone 5 | -0.17 (0.13) | -0.32 (0.12) | -0.31 (0.13)
  Zone 6 | 0.00 (0.14) | -0.02 (0.13) | -0.15 (0.14)

7. Secondary Outcome: Conjunctival Hyperemia Grading
Description: Mean change from baseline in zonal conjunctival hyperemia in study eye using a 0- to 4-unit clinical grading scale and standardized grading photos, with 0 being better and 4 being worse
Time Frame: 8 weeks
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
units on a scale
  Frontal | -0.17 (0.07) | -0.15 (0.07) | -0.13 (0.07)
  Nasal | -0.20 (0.07) | -0.13 (0.07) | -0.24 (0.07)
  Temporal | -0.18 (0.08) | -0.08 (0.08) | -0.21 (0.08)

8. Secondary Outcome: Tear Film Break-up Time (TBUT)
Description: Mean change from baseline in TBUT in study eye
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
seconds | 0.29 (0.26) | 0.13 (0.25) | 0.18 (0.26)

9. Secondary Outcome: Schirmer's Test
Description: Mean change from baseline in tear volume in study eye as assessed by unanesthetized Schirmer test
Time Frame: 8 weeks
Population: PP Population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
Number analyzed (Participants) | 46 | 46 | 46
mm | 1.64 (0.94) | 1.92 (0.91) | 2.50 (0.93)

ADVERSE EVENTS:
Time Frame: Duration of study (8 weeks)
Arm/Group | Vehicle Ophthalmic Solution | ALY688 Ophthalmic Solution 0.1% | ALY688 Ophthalmic Solution 0.4%
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 1/46 | 0/46
Other Adverse Events (participants affected / at risk) | 9/46 | 6/46 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Ophthalmic Solution (N=46) | ALY688 Ophthalmic Solution 0.1% (N=46) | ALY688 Ophthalmic Solution 0.4% (N=46)
vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Ophthalmic Solution (N=46) | ALY688 Ophthalmic Solution 0.1% (N=46) | ALY688 Ophthalmic Solution 0.4% (N=46)
Instillation site pain (General disorders) | 9 (18) | 6 (12) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT04201574/Prot_SAP_001.pdf